CLINICAL TRIAL: NCT04566159
Title: Computer Delivered and Community Health Worker Supported Smoking Cessation Intervention for Hospitalized Persons With HIV
Brief Title: Computer Delivered and Community Health Worker Supported Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00117151-2
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Smoking
Keywords: HIV
MeSH Terms: conditions — Tobacco Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBI + CHW (Experimental): 2 Session Computer Delivered Intervention with use of Nicotine Replacement Therapy and Community Health Worker Follow Up
  Interventions: Behavioral: CBI-CHW
- Routine Care (Other): Routine Tobacco Cessation Advice to Stop Smoking and Nicotine Replacement Therapy as offered by the inpatient team
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: CBI-CHW — 2 sessions of computer delivered counseling + nicotine replacement therapy and CHW follow up post hospitalization up to twice weekly for up to 8 weeks
  Arms: CBI + CHW
Other: Standard Care — Standard tobacco treatment care offered by the inpatient care
  Arms: Routine Care

SUMMARY:
The prevalence of tobacco smoking is high among persons with HIV (PWH). The investigators are piloting a two session computer-delivered intervention (CBI) with linkage to a community health worker (CHW) among hospitalized PWH with tobacco use 1a) To determine feasibility and acceptability of delivering this intervention and 2a) To determine intervention effect on 1) readiness to quit smoking and confidence in ability to quit smoking 2) uptake of smoking cessation therapy

ELIGIBILITY:
Inclusion Criteria:

* Age >=18,
* A patient admitted to the Johns Hopkins Hospital
* Smoked >100 cigarettes in their lifetime
* Current smoker
* English speaking

Exclusion Criteria:

* Contraindication to nicotine replacement therapy including unstable angina and acute coronary syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility as assessed by the Feasibility of Intervention Measure | 3 months
  4 item scale, maximum score of 20 with higher score indicating greater feasibility
Intervention Acceptability as assessed by the Acceptability of an Intervention Measure | 3 months
  Noted as continuous score on 4 item scale, maximum value of 20 with higher score indicating greater acceptability

SECONDARY OUTCOMES:
Readiness to quit smoking as assessed by a Visual analog scale | immediately post intervention
  Score of 10=Ready to Quit, Score of 1=Not ready to quit. Scale is from 1-10
Uptake of nicotine replacement therapy | immediately post intervention
  Dichotomous yes/no.
Continued use of nicotine replacement therapy 1 month post intervention | 30 days post intervention
  Dichotomous yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
As this is a very small pilot, we will share de-identified data on request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion
Access Criteria: Information will be shared on request. Requests can be made to the study PI who will then work with the data manager to compile a de-identified data set.